CLINICAL TRIAL: NCT06541886
Title: Adapted CBT-I for Adolescents With Insomnia : The DREAM-IT Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: American Academy of Sleep Medicine (Other); Nyxeos Consulting (Unknown)
Responsible Party: Principal Investigator, Sarah Honaker, Associate Professor of Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13047; 249-SR-21 (Other Grant/Funding Number: American Academy of Sleep Medicine Foundation)
Record Dates: First submitted 2024-07-23; First posted 2024-08-07 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Insomnia
Keywords: Cognitive Behavioral Therapy for Insomnia; Adolescence; Randomized controlled trial; Efficacy; Stakeholders; Adaptation; Actigraphy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: This study has a parallel intervention study model. Participants are assigned to one of two groups in parallel for the duration of the study-either Teen CBT-I or waitlist control for 8 weeks.
Masking Description: Participants assigned to either condition will know about their assignment as they either will or will not receive treatment with a therapist during the 8-week active treatment period. Care providers, investigators, and outcome assessors will also be aware of group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Teen CBT-I (Experimental): Teens in this treatment condition will have an intake session and 6 treatment sessions virtually and individually with a therapist. The first session will include an introduction to Sleep Science and Insomnia Treatment. Middle sessions will include Healthy Sleep Habits, Setting a Sleep Schedule, Preparing the Mind and Body for Sleep, and Distinguishing the Sleep Space and Wake Space. The final session will be be centered on maintenance of treatment gains. Treatment will also include visual aids (e.g., slides) to convey didactic or psychoeducational material.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I)
- Waitlist (No Intervention): Teens in the waitlist condition will still complete the same study measures and receive the same payment for taking part in the study, but they will not receive treatment from a therapist. Their treatment will begin after they have completed the second round of measures (i.e., 8 weeks after they complete the baseline assessment). After they have completed the second round of measures, they will be given free access to an app that provides guided insomnia treatment. While no live therapist is involved, the approach is similar to traditional CBT-I.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia (CBT-I) — CBT-I was developed as a treatment for adults with insomnia. There are more than 100 studies showing that CBT-I is effective in treating insomnia in adults, and several studies suggest it is also effective in treating insomnia in teens.
  Arms: Teen CBT-I

SUMMARY:
The goal of this study is to test an adapted treatment for teen insomnia in comparison to a waitlist condition. Cognitive Behavioral Therapy for Insomnia (CBT-I) is an intervention that was developed for adults and is sometimes also used for teens. Teens, parents, and health care providers helped to review and adapt CBT-I to form Teen CBT-I. Teen CBT-I includes most of the same content as CBT-I, with some changes to match teen biology and lifestyles.

The main questions this clinical trial aims to answer are:

* Does Teen CBT-I improve insomnia symptoms in teens?

  o Researchers will compare Teen CBT-I to the waitlist control condition to see if insomnia symptoms significantly improve in the treatment group.
* Do teens and their parents find Teen CBT-I to be acceptable? o Researchers will examine Teen CBT-I acceptability ratings.

Teen CBT-I is hypothesized to improve insomnia symptoms in teens, and teens and parents are hypothesized to find Teen CBT-I to be acceptable.

Teen participants will be randomized to one of the two conditions: Teen CBT-I treatment or waitlist control. They will also complete assessments at three timepoints: Baseline (before treatment); post-intervention (after treatment); and follow-up (2 months after treatment). For each assessment, teen participants will:

* Fill out questionnaires about their sleep, mood, and other areas
* Keep daily sleep logs for one week
* Wear an actigraph, a wrist-watch like device that records activity levels to determine sleep-wake patterns, for one week.

Parent participants will also be asked to complete questionnaires at each measurement point about their teen's sleep, mood, and other areas.

The intervention conditions are:

* Teen CBT-I includes 4-6 one-hour individual virtual sessions with a therapist. It includes standard CBT-I content with some small changes to match teen biology and lifestyles. The main parts of this treatment include healthy sleep habits, only using the bed for sleep, keeping a recommended sleep schedule, changing negative thoughts about sleep, and learning ways to relax the mind and body for sleep.
* Waitlist-control, in which teens will not receive any treatment for 8 weeks. After the second assessment, they will receive free access to an app-based CBT-I treatment which they can complete on their own.

DETAILED DESCRIPTION:
Background: Cognitive Behavioral Therapy for Insomnia (CBT-I) has been well-established as an efficacious and first-line treatment for insomnia in adults, but research on its use with adolescents is limited. Preliminary evidence for the efficacy of CBT-I with adolescents is promising, but treatment protocols in existing trials are heterogeneous, making it difficult to characterize CBT-I for teens. In Aim 1 of this study, CBT-I was systematically adapted through collaboration with stakeholders (i.e., teens, parents, and behavioral sleep medicine providers across the country), making changes to the intervention tailored to teen biology and lifestyles.

Objective: The objective of this study is to test this adapted intervention (hereafter referred to as Teen CBT-I) in comparison to a waitlist control condition in adolescents with insomnia.

Hypotheses:

1. Teen CBT-I will reduce insomnia symptoms compared to a no treatment (waitlist) condition.
2. Teen CBT-I will be deemed acceptable by teens and parents.

Participants: Adolescents with insomnia (N=28) and their parents will be randomized to either Teen CBT-I (n=14) or the waitlist control condition (n = 14).

Recruitment: Parents of adolescents will be recruited via social media. Recruitment posts and images will be boosted to both Facebook and Instagram using the Facebook Ads Manager system. Recruitment posts and images will briefly describe the study and provide a link to an Interest Survey for parents to complete. Parents can then provide consent and contact information for their teen to also be contacted and invited to complete a recruitment survey.

Interest Survey:

The online surveys will provide additional information about the study and ask eligibility questions. Ineligible respondents will be informed of their status and will not be asked for any additional information. Respondents who are not ineligible* will be asked for contact information and demographic information.

Some, but not all, interested participants will be contacted and invited to complete the next step, an Eligibility and Consent Meeting.

*Some eligibility criteria will be assessed during the Eligibility and Consent meeting as they are more complex and require evaluation through an interactive call rather than a survey.

Eligibility and Consent Meeting:

Parent-teen dyads who completed the recruitment surveys and are not screened out will then be asked to meet with a research team member to further determine eligibility. Teen suicidal ideation will be evaluated, along with other comorbid conditions that may make the teen ineligible.

If the teen and parent are determined to be eligible for the study, an informed consent process will then be initiated. Parents and teens will be provided with more information about the study and the opportunity to ask questions, prior to deciding whether or not they would like to be part of the study. Enrolled participants will then proceed to the baseline assessment.

Randomization Once the baseline measures are completed, the teen-parent dyad will be randomized to one of the two conditions using a randomization module in REDCap. Randomization will be stratified based on age so that there is the same number of younger teens (ages 13-15) and older teens (ages 16-18) in each condition.

Conditions Participants randomized to Teen CBT-I will meet individually with a therapist for a virtual, one-hour session. Each session will be administered free of charge. Most of each treatment session will be with just the therapist and the teen. However, the parent will be asked to join for the last ten minutes of each appointment to keep the parent informed about the treatment plan. If they wish, teens can decide to involve their parent earlier in the session.

Teen CBT-I Teens in this treatment condition will have an intake session and between 4 to 6 treatment sessions. The first session will include an introduction to sleep science and insomnia treatment. Middle sessions will include Healthy sleep habits, Setting a sleep schedule, Preparing the mind and body for sleep, and Distinguishing the sleep space from the teen's hang out space. The last session will be centered on maintenance of treatment gains. Treatment will include visual aids (e.g., a powerpoint) to convey didactic or psychoeducational material.

Waitlist Control Teens in the waitlist condition will still complete the same study measures, but they will not receive treatment from a therapist. Their treatment will begin after they have completed the second round of measures (i.e., 8 weeks after completing the baseline measures). After they have completed the second round of measures, they will be given free access to an app that provides guided insomnia treatment. While no live therapist is involved, the approach is similar to traditional CBT-I.

Fidelity Monitoring Audio and video will be recorded during the treatment sessions. The purpose of this is so that supervisors can review some of the sessions to help with therapist training, and to make sure that the therapist is following the treatment protocol. These recordings will only be reviewed by the study team to monitor the therapist, and recordings will be stored securely. No one outside of the study will have access to these recordings. The recordings will be deleted after the 2-month follow up. De-identified (i.e., without names, location) transcripts of the sessions will be kept. If a teen-parent dyad is not comfortable with recording of the sessions, they can opt out, meaning that they can still be in the study, but their treatment sessions will not be recorded. There is an opt-in / opt-out component within the informed consent process.

Analysis Plan Linear regression modeling will be used to assess pre- and post-intervention changes in clinical outcomes, reporting effect sizes (Cohen's d) and controlling for relevant covariates.

Implementation outcomes will be reported descriptively. With n=28 (comparing two groups in multiple pairwise comparisons), 80% power, and α = .05, there is adequate power to detect an effect size of d = 1.00, which is consistent with prior research testing CBT-I for teens and adults, with effect sizes ranging from d = 1.00-1.22.

Potential Risks Potential risks include confidentiality breaches and discomfort from wearing the actigraph, a wrist-watch like device that will be used to measure adolescent sleep outcomes.

The risk of loss of confidentiality will be minimized by the research team. Efforts will be made to keep personal information confidential, and only de-identified group data will be shared or published to keep participant identity confidential. Personal information would only be disclosed if required by law.

Completed questionnaires will be stored in a secure, electronic database that is accessible only by study team members approved by the Office for Protection of Human Subjects.

One exception to confidentiality would be if there is concern about the health and safety of a teen. This risk would be immediately discussed with the teen and parent and reported to the necessary authorities to ensure safety. An example of this would be if a teen indicated they were being abused or that they were planning to hurt themselves or someone else.

Another exception to confidentiality is that the university and federal offices that are in charge of protecting the rights of research participants and the quality of research may, in rare instances, need to inspect or copy a researcher's data. This includes the Indiana University Institutional Review Board and the Office for Human Research Protections.

Although extremely rare, if a participant experiences skin discomfort from the actigraph, they can wear the device over a shirt.

It is also possible that participants could lose or damage the actigraph. Research staff will explain the proper use and importance of these devices to prevent such risks, but the risk is still possible. If a participant loses or damages the actigraph, they will not be held financially responsible and will not be excluded from the study. Data within the actigraph can only be accessed with specialized software. In addition, no identifiers are included in the actigraphic output aside from the participant's research ID.

Informed consent. The process will be conducted in a location that is considered private and controlled. The consenting process will include the study purpose, inclusion/exclusion criteria, enrollment goal, timeline and study interventions. The adolescent participant will assent for the study following IRB guidelines along with obtaining consent from adult participants. All participants will be asked to provide verbal consent/assent prior to participation in any study activities or interventions.

Potential benefits of the proposed research to human subjects and others Benefits to participants may include improvement in insomnia symptoms. The potential benefit to society is determining whether the adapted treatment protocol is efficacious. If it is, it can then be used more widely to improve outcomes for adolescents with insomnia. This can lead to improved functioning in adolescents with insomnia and intervention success for providers and caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents (13-18 years) who are in either middle school or high school and meet ICSD-3 diagnostic criteria for Chronic Insomnia Disorder, currently or in the past year, based on self-reported insomnia symptoms, using a screening checklist.
* Reside in a state where Dr. McQuillan (supervising provider) is licensed to practice psychology (with PsyPact) which are the following states: Alabama, Arizona, Arkansas, Colorado, Commonwealth of the Northern Mariana Islands, Connecticut, Delaware, District of Columbia, Florida, Georgia, Idaho, Illinois, Indiana, Kentucky, Maine, Maryland, Michigan, Minnesota, Mississippi, Missouri, Nebraska, Nevada, New Hampshire, New Jersey, North Carolina, North Dakota, Ohio, Oklahoma, Pennsylvania, Rhode Island, South Carolina, South Dakota, Tennessee, Texas, Utah, Vermont, Virginia, Washington, West Virginia, Wisconsin, and Wyoming.
* Sufficient English language proficiency for consent and study participation
* Reliable internet access to attend virtual visits with audio and video
* Parents or other caregivers of these adolescents (hereafter referred to as a parent) must live in the home with the identified adolescent at least 50% of the time and must report playing a parental role for that adolescent. The parent must also be able to attend the final 10 minutes of each treatment session, if the teen is randomized to a treatment condition.

Exclusion Criteria:

* Sleep aid use that is either inconsistent (e.g., used some but not all nights) and cannot be discontinued OR consistent and effective enough that the teen no longer has insomnia symptoms while using it. If a teen agrees to keep the dose and frequency of sleep aid use consistent throughout the treatment and still has insomnia symptoms at baseline, they are not ineligible.
* Prior participation in Aim 1 of DREAM IT study (e.g., participation in an Aim 1 focus group).
* Comorbid medical or psychiatric conditions, including substance use disorders, that are acute, unstable, or untreated. Individuals with Autism Spectrum Disorder, Epilepsy, Schizophrenia, and Bipolar Disorder will be excluded.
* Comorbid delayed sleep wake phase disorder or other active/untreated sleep disorders, including RLS, OSA, and Nightmare disorder
* Active suicidal ideation with plan and intent

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Teen-reported insomnia severity | Baseline, Post-treatment (approximately 8 weeks after baseline), and 2 month follow up
  assessed via the PROMIS (Patient-Reported Outcomes Measurement Information System) sleep disturbance scale, which has been established as reliable and valid with adolescents. Possible scores on this scale range from 10 - 50, where higher scores reflect more severe insomnia.
Teen-reported treatment acceptability | Post-treatment (approximately 8 weeks after baseline)
  based on the widely used Client Satisfaction Questionnaire, which assesses treatment feasibility, satisfaction, and perceived helpfulness. Possible scores on this scale range from 8-40, where higher scores reflect higher acceptability ratings.

SECONDARY OUTCOMES:
Teen-reported sleep onset latency | Baseline, Post-treatment (approximately 8 weeks after baseline), and at 2-month follow up
  Based on sleep diary
Teen-reported wake after sleep onset | assessed at Baseline, Post-treatment (approximately 8 weeks after baseline), and at 2-month follow up
  Based on sleep diary
Teen-reported night wakings | assessed at Baseline, Post-treatment (approximately 8 weeks after baseline), and at 2-month follow up
  Number of night wakings, based on sleep diary
Teen-reported sleep efficiency | assessed at Baseline, Post-treatment (approximately 8 weeks after baseline), and at 2-month follow up
  Average of total sleep time divided by time spent in bed each night, based on information provided by teen in the sleep diary
Sleep efficiency | assessed at Baseline and Post-treatment (approximately 8 weeks after baseline)
  Average of total sleep time divided by time spent in bed each night, as measured via the actigraph
Wake after sleep onset | assessed at Baseline and post-treatment (approximately 8 weeks after baseline)
  Based on actigraphy
Teen Mood | assessed at Baseline, Post-treatment (approximately 8 weeks after baseline), and at 2-month follow up
  Depressive Symptoms from the PROMIS (Patient-Reported Outcomes Measurement Information System) measure. Possible scores range from 8 to 40, where higher scores reflect more depressive symptoms.
Teen Stress | assessed at Baseline, Post-treatment (approximately 8 weeks after baseline), and at 2-month follow up
  Teen report on the PROMIS (Patient-Reported Outcomes Measurement Information System) Psychological Stress Experiences measure. Possible scores range from 8 to 40, where higher scores reflect more stress.
Teen Daytime Sleepiness | assessed at Baseline, Post-treatment (approximately 8 weeks after baseline), and at 2-month follow up
  Teen report on the PROMIS (Patient-Reported Outcomes Measurement Information System) Sleep-Related Impairment Scale. Possible scores range from 8 to 40, where higher scores reflect more daytime impairment.
Teen-reported sleep hygiene | assessed at Baseline, Post-treatment (approximately 8 weeks after baseline), and at 2-month follow up
  pediatric sleep practices questionnaire - short form. Possible scores range from 7 to 35, where higher scores reflect better sleep hygiene.
Teen-reported parent-teen conflict about sleep | assessed at Baseline, Post-treatment (approximately 8 weeks after baseline), and at 2-month follow up
  "How much did you and your parent argue about sleep in the past week ?" Using a 1-5 Likert scale, where higher scores reflect more conflict.
Parent-reported parent-teen conflict about sleep | assessed at Baseline, Post-treatment (approximately 8 weeks after baseline), and at 2-month follow up
  "How much did you and your teen argue about sleep in the past week ?" Using a 1-5 Likert scale, where higher scores reflect more conflict.
Parent-reported insomnia symptoms | assessed at Baseline, Post-treatment (approximately 8 weeks after baseline), and at 2-month follow up
  using the parent-report PROMIS (Patient-Reported Outcomes Measurement Information System) sleep disturbance scale. Possible scores range from 10 - 50, where higher scores reflect more severe insomnia.
Parent-reported daytime sleepiness | assessed at Baseline, Post-treatment (approximately 8 weeks after baseline), and at 2-month follow up
  using the parent-report PROMIS (Patient-Reported Outcomes Measurement Information System) sleep related impairment scale. Possible scores range from 8 to 40, where higher scores reflect more severe daytime impairment.
Parent perception of adolescent mood | assessed at Baseline, Post-treatment (approximately 8 weeks after baseline), and at 2-month follow up
  using the parent-report PROMIS (Patient-Reported Outcomes Measurement Information System) depressive symptoms scale. Possible scores range from 6 to 30, where higher scores reflect more teen depressive symptoms.
Parent-reported school attendance | assessed at Baseline, Post-treatment (approximately 8 weeks after baseline), and at 2-month follow up
  Based on two items: "In the past 2 weeks, how many days has your child missed school because of difficulty sleeping?" AND "In the past 2 weeks, how many days has your child been late to school because of difficulty sleeping?"
Teen-reported treatment adherence | assessed at Post-treatment (approximately 8 weeks after baseline) and at 2-month follow up
  via adolescent report on sleep diary
Treatment engagement | assessed at post-treatment approximately 8 weeks after baseline
  based on session attendance and treatment completion
Adverse treatment effects | assessed at post-treatment approximately 8 weeks after baseline
  Report of any car accidents, suicidality, or risky behaviors that could be attributed to sleep restriction and/or reductions in daytime alertness
Parent-reported treatment acceptability | assessed at post-treatment approximately 8 weeks after baseline
  based on the widely used Client Satisfaction Questionnaire, which assesses treatment feasibility, satisfaction, and perceived helpfulness. Possible scores on this scale range from 8-40, where higher scores reflect higher acceptability ratings.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah M Honaker, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No